CLINICAL TRIAL: NCT02584582
Title: The Effect of GLP-1 on Postprandial Glucagon Secretion During Prolonged and Intermittent Stimulation of the GLP-1 Receptor Independent of The Gastric Emptying Rate. A Randomized, Open-label Study in People With Type 1 Diabetes
Brief Title: The Effect of GLP-1 on Postprandial Glucagon Secretion Independent of The Gastric Emptying Rate
Acronym: ALFA-1
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Christan SS Frandsen, MD, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-3-2014-128
Record Dates: First submitted 2015-08-06; First posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Type 1 Diabetes
Keywords: Glucagon; Glukagon-like peptide-1 (GLP-1); GLP-1 receptor agonist (GLP-1RA); Incretins
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Liraglutide; Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Liraglutide + Liquid meal test (Experimental): Liraglutide 1.2 mg once daily for 14 days (0.6 mg/day for one week, escalated to 1.2 mg/day after one week)
  Interventions: Drug: Liraglutide; Procedure: Liquid meal test
- Exenatide + Liquid meal test (Experimental): Exenatide 10 mcg twice daily for 14 days (5 mcg twice daily for one week, escalated to 10 mcg twice daily after one week)
  Interventions: Drug: Exenatide; Procedure: Liquid meal test
- Baseline + Liquid meal test (Other): Baseline day with no additional medication
  Interventions: Procedure: Liquid meal test; Other: No drug (Baseline day)

INTERVENTIONS:
Drug: Liraglutide
  Arms: Liraglutide + Liquid meal test
Drug: Exenatide
  Arms: Exenatide + Liquid meal test
Procedure: Liquid meal test
Other: No drug (Baseline day)
  Arms: Baseline + Liquid meal test

SUMMARY:
Aim: To investigate the glucagonostatic effect of glucagon-like peptide-1 (GLP-1) independent of the gastric emptying rate.

DETAILED DESCRIPTION:
Aim: To investigate the glucagonostatic effects of glucagon-like peptide-1 (GLP-1) during prolonged and intermittent stimulation of the GLP-1 receptor independent of the gastric emptying rate. Glucagon concentrations will be measured following a liquid meal administered in duodenum at baseline and after exenatide, and liraglutide treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes
* >18 years
* No residual beta-cell function (stimulated C-peptide < 60 pmol)

Exclusion Criteria:

* Pancreatitis
* gastroparesis
* history of alcohol and/or drug abuse
* pregnancy and lactation
* other medical or psychological condition that made the patient unsuitable for study participation according to the investigators´ assessment
* contraindications to gastroscopy
* cancer (unless in complete remission > five years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Glucagon concentration (postprandial) | 4 hours
  glucagon area under the curve (AUC) (0-240 minutes) and baseline to peak increments will be calculated

SECONDARY OUTCOMES:
Postprandial glucose concentrations | 4 hours
  glucose AUC (0-240 minutes) and baseline to peak increments will be calculated
glucagon-like peptide-1 (GLP-1) | 4 hours
  GLP-1 AUC (0-240 minutes) and baseline to peak increments will be calculated
glucagon-like peptide-2 (GLP-2) | 4 hours
  GLP-2 AUC (0-240 minutes) and baseline to peak increments will be calculated
glucose-dependent insulinotropic polypeptide (GIP) | 4 hours
  GIP AUC (0-240 minutes) and baseline to peak increments will be calculated
Cholecystokinin (CCK) | 4 hours
  CCKAUC (0-240 minutes) and baseline to peak increments will be calculated
Peptide YY (PYY) | 4 hours
  PYY AUC (0-240 minutes) and baseline to peak increments will be calculated
Ghrelin | 4 hours
  Ghrelin AUC (0-240 minutes) and baseline to peak increments will be calculated
Gastrin | 4 hours
  Gastrin AUC (0-240 minutes) and baseline to peak increments will be calculated
Oxyntomodulin | 4 hours
  Oxyntomodulin AUC (0-240 minutes) and baseline to peak increments will be calculated
Free fatty acids (FFA) | 4 hours
  FFA AUC (0-240 minutes) and baseline to peak increments will be calculated
triacylglycerol (TAG) | 4 hours
  TAG AUC (0-240 minutes) and baseline to peak increments will be calculated